CLINICAL TRIAL: NCT01718964
Title: Acute Effects of Cortisol on Heroin Craving in Opioid Dependence
Brief Title: Acute Effects of Cortisol on Heroin Craving in Opioid Dependence (Ghost-Basel)
Acronym: Ghost-Basel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dominique de Quervain, MD (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Professor MD, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012DR2144
Record Dates: First submitted 2012-10-23; First posted 2012-11-01 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Hydrocortisone; Mannitol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Other): Cortisol 20 mg /Placebo Mannitol
  Interventions: Drug: Cortisol 20 mg; Drug: Mannitol
- B (Other): Placebo Mannitol/Cortisol 20mg
  Interventions: Drug: Cortisol 20 mg; Drug: Mannitol

INTERVENTIONS:
Drug: Cortisol 20 mg
Drug: Mannitol — Mannitol used as placebo

SUMMARY:
To investigate the effects of cortisol on heroin craving and stress reaction in heroin addicted subjects Randomized, double-blind, placebo-controlled, cross-over, single administration of study medication Study hypothesis:Cortisol has an inhibiting effect on heroin craving and stress reactivity in opioid dependent subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Opioid dependency
* Participant in the Janus heroin programme of the UPK Basel
* Able to control parallel consumption of other drugs
* Stable i.v. substitution for at least 3 months

Exclusion Criteria:

* co-morbid psychiatric disturbances
* Current medical conditions excluding participation
* Recent history of systemic or topic glucocorticoid therapy
* known hypersensitivity to the IMP under investigation (cor-tisol)
* pregnancy, breast-feeding
* inability to read and understand the participant's information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Heroin craving | baseline, change from baseline during and after presentation of drug stimuli
  outcome measures will be taken during the participants 2 test visit days. Each participant will stay for approx. 3 hours.

SECONDARY OUTCOMES:
Anxiety | baseline, change from baseline during and after presentation of drug stimuli
  outcome measures will be taken during the participants 2 test visit days. Each participant will stay for approx. 3 hours.

OTHER OUTCOMES:
Symptoms of withdrawal | baseline, change from baseline during and after presentation of drug stimuli
  outcome measures will be taken during the participants 2 test visit days. Each participant will stay for approx. 3 hours.
saliva cortisol level | baseline, change from baseline during and after presentation of drug stimuli
  outcome measures will be taken during the participants 2 test visit days. Each participant will stay for approx. 3 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric Hospital, Basel, Switzerland

REFERENCES:
- [Derived] Walter M, Bentz D, Schicktanz N, Milnik A, Aerni A, Gerhards C, Schwegler K, Vogel M, Blum J, Schmid O, Roozendaal B, Lang UE, Borgwardt S, de Quervain D. Effects of cortisol administration on craving in heroin addicts. Transl Psychiatry. 2015 Jul 28;5(7):e610. doi: 10.1038/tp.2015.101. PMID 26218852